CLINICAL TRIAL: NCT03419819
Title: Evaluation of the Acceptability, Tolerance, and Satiety of PKU Sphere, a Glycomacropeptide (GMP) Based Medical Food in Patients With Phenylketonuria (PKU).
Brief Title: Evaluation of PKU Sphere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT-PKUS-2016-11-28
Record Dates: First submitted 2018-01-03; First posted 2018-02-05 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonurias
Keywords: Phenylketonuria; GMP; Sphere; Child; Adult; Phenylalanine; PKU; Glycomacropeptide
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Two phase study consisting of a 1 week taste introduction period followed by a 4 week period assessing acceptability and metabolic control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU Sphere (Experimental): Phase 1: 1 week To evaluate the acceptability of PKU Sphere during a short-term (1 week) period. Individuals with PKU will aim to consume a minimum of 30% of the medical food component of the diet as PKU Sphere. The amount will be assessed and advised on an individual basis.
  Phase 2: 4 weeks To evaluate longer-term acceptability and metabolic control in individuals with PKU consuming an agreed target of 50 - 100% of their medical food component of the diet as PKU Sphere for 4 weeks. Some individuals, particularly young children between the ages of 3 - 6 years, may require a 1 - 3 week build up period to reach target volume which will be assessed on an individual basis.
  Interventions: Dietary Supplement: PKU Sphere

INTERVENTIONS:
Dietary Supplement: PKU Sphere — PKU Sphere is a glycomacropeptide based alternative to amino-acid based products for the dietary management of phenylketonuria.

SUMMARY:
A prospective, open-label study of PKU Sphere in patients with PKU following a phenylalanine restricted therapeutic diet.

DETAILED DESCRIPTION:
The rationale for this study is to assess acceptability, adherence and metabolic control in individuals with PKU consuming PKU Sphere, a GMP-based medical food.

The sponsor developed PKU Sphere in response to growing interest in GMP medical foods for the purpose of improving adherence and quality of life by offering an alternative to amino acid based medical foods. PKU Sphere is a powdered, low phenylalanine medical food containing a balanced mix of casein glycomacropeptide (GMP) isolate, essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals and the long chain polyunsaturated fatty acid (LCP); docosahexaenoic acid (DHA). PKU Sphere has been designed for use in the dietary management of Phenylketonuria. It is available in two flavors, Red Berry and Vanilla, packaged in individual serving sachets of 35g and containing 20g protein equivalent (PE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU, identified by newborn screening (NBS) and treated since birth.
* Ages 3 years and above (this includes pregnant women who will be assessed on an individual basis by the Co-Principal Investigators).
* Currently or previously consuming a low phenylalanine diet supplemented with a medical food designed for the dietary management of PKU.
* English as primary language.
* Willingly given, written, informed consent from the participant, 18 or more years, or from the parent/caregiver for participants < 18 years.
* Willingly given, written assent (if appropriate) for those < 18 years.

Exclusion Criteria:

* Currently consuming 100% of the medical food component of the diet as PKU sphere.
* An inability, in the opinion of the investigator, to comply with the requirements of the protocol.
* Any other type of inherited metabolic disease.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Phase 1: taste | Days 1 - 7.
  Questionnaire data captured to evaluate taste
Phase 1: smell | Days 1 - 7.
  Questionnaire data captured to evaluate smell
Phase 1: texture | Days 1 - 7.
  Questionnaire data captured to evaluate texture
Phase 1: gastrointestinal tolerance | Days 1 - 7.
  Questionnaires will be completed daily during the 1-week taste test.
Phase 1: phenylalanine concentration | Days 1 and 7.
  Phenylalanine concentrations measured via blood spot analysis.
Phase 1: tyrosine concentration | Days 1 and 7.
  Tyrosine concentrations measured via blood spot analysis.
Phase 2: quantitative change in plasma amino acids at day 28 | Phase 2, day 1 and day 28.
  Compare comprehensive plasma amino acid profiles at baseline and end of the trial.
Phase 2: gastrointestinal tolerance | Phase 2, days 1 - 28.
  Questionnaires will be completed daily throughout Phase 2.
Phase 2: change in 3-day diet record at end of study | Phase 2, days 1 - 3 and days 26 - 28.
  A 3-day diet record will be completed in the first 3 days and the last 3 days for comparison.
Phase 2: change in anthropometry at end of study | Phase 2, days 1 and 28.
  Participants will be weighed and measured, a growth chart plotted (children only), and BMI calculated
Phase 2: phenylalanine concentration | Twice weekly for four weeks during phase 2
  Phenylalanine concentrations measured via blood spot analysis.
Phase 2: tyrosine concentration | Twice weekly for four weeks during phase 2
  Tyrosine concentrations measured via blood spot analysis.
Phase 2: questionnaire data captured to evaluate change in taste perception | Phase 2, days 14 and 28.
  Data captured to evaluate taste
Phase 2: questionnaire data captured to evaluate change in smell perception | Phase 2, days 14 and 28.
  Data captured to evaluate smell
Phase 2: questionnaire data captured to evaluate change in texture perception | Phase 2, days 14 and 28.
  Data captured to evaluate texture

SECONDARY OUTCOMES:
Phase 1: questoinnaire evaluating subjective measures of satiety | Phase 1, days 1 - 7.
  To evaluate if PKU Sphere increases subjective measures of satiety
Phase 2: questoinnaire evaluating subjective measures of satiety | Phase 2, days 1, 14 and 28.
  To evaluate if PKU Sphere increases subjective measures of satiety

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Van Calcar, PhD, Principal Investigator — Oregon Health and Science University; Joyanna Hansen, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No